CLINICAL TRIAL: NCT00312013
Title: A Randomized, Controlled Trial to Evaluate the Effects of Nadroparin on Survival and Disease Progression in Patients With Advanced Malignancies of the Lung, Pancreas, or Prostate
Brief Title: Effects Of Nadroparin In Patients With Lung, Pancreas Or Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FRX106365
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Thrombosis, Venous
Keywords: low molecular weight heparin; nadroparin; non-small cell lung cancer; cancer survival; prostate cancer; pancreatic cancer
MeSH Terms: conditions — Venous Thrombosis; Carcinoma, Non-Small-Cell Lung; Prostatic Neoplasms; Pancreatic Neoplasms | interventions — Nadroparin

ARMS (2):
- No Nadroparin (No Intervention): Patients will receive all standard anticancer treatment. Patients in this arm will not receive nadroparin
- Nadroparin (Experimental): Patients will be randomized to receive standard anticancer treatment. Nadroparin patients will be treated with therapeutic doses of subcutaneous (s.c). nadroparin for 2 weeks followed by half therapeutic doses for 4 weeks. After 4 weeks of wash-out, subsequent 2-week periods of therapeutic doses of nadroparin will be given for a total of 6 cycles each separated by a 4-week wash-out. The study treatment period ends at week 46 regardless of number of cycles achieved at that moment.
  Interventions: Drug: Nadroparin

INTERVENTIONS:
Drug: Nadroparin — Patients will received all standard anti-cancer treatments. Therapeutic doses of nadroparin will be administered, subcutaneous for 2 weeks followed by half therapeutic doses for 4 weeks. After 4 weeks of wash-out, subsequent 2 week periods of therapeutic doses will be given for a total of 6 cycles each separated by a 4 week wash out. The study treatment period ends at week 46 regardless of the number of cycles achieved.
  Arms: Nadroparin

SUMMARY:
This study will evaluate the effects of nadroparin on survival and disease progression in patients with hormone-refractory prostate cancer (HRPC), locally advanced pancreatic cancer or non-small-cell lung carcinoma (NSCLC).

ELIGIBILITY:
Inclusion criteria:

* Hormone refractory prostate cancer within 6 months of diagnosis, OR locally advanced (non-metastasized) pancreatic cancer within 3 months of diagnosis, OR non-small-cell lung cancer within 3 months of stage IIIB.

Exclusion criteria:

* Life expectancy of <3 months.
* Poor performance status (Karnofsky <60).
* Need to be on anticoagulants.
* Use of nadroparin (a low molecular weight heparin) for any reason including a history of heparin-induced thrombocytopenia.
* Have brain metastasis.
* At a high risk of bleeding or have a platelet count <50,000/mm3.
* Have very poor kidney function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2006-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Death due to all causes at study end (patients will be followed until at least Week 46 after randomization). | AT least 46 weeks after randomization

SECONDARY OUTCOMES:
Time to tumor progression | 46 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (80):
- Belgium (6):
  - GSK Investigational Site, Aalst
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Brasschaat
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Roeselare
- GSK Investigational Site, Toronto, Ontario, Canada
- Czechia (3):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Příbram
- France (9):
  - GSK Investigational Site, Béthune
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pierre-Bénite
  - GSK Investigational Site, Saint-Priest-en-Jarez
  - GSK Investigational Site, Strasbourg
- Germany (21):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Ebensfeld, Bavaria
  - GSK Investigational Site, Planegg, Bavaria
  - GSK Investigational Site, Bremen, City state Bremen
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Fulda, Hesse
  - GSK Investigational Site, Giessen, Hesse
  - GSK Investigational Site, Greifenstein, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Herne, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Bad Berka, Thuringia
- Hungary (3):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Győr
  - GSK Investigational Site, Törökbálint
- Italy (8):
  - GSK Investigational Site, Chieti Scalo, Abruzzo
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Bergamo, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Campobasso, Molise
  - GSK Investigational Site, Florence, Tuscany
  - GSK Investigational Site, Padua, Veneto
- Netherlands (13):
  - GSK Investigational Site, Almelo
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Delft
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Nieuwegein
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Sittard
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Winterswijk
  - GSK Investigational Site, Zwolle
- Poland (5):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lubin
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Warsaw
- Russia (9):
  - GSK Investigational Site, Arkhangelsk
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Kirov
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Omsk
  - GSK Investigational Site, Orenburg
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Voronezh
- Slovenia (2):
  - GSK Investigational Site, Golnik
  - GSK Investigational Site, Ljubljana

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] van Doormaal FF, Di Nisio M, Otten HM, Richel DJ, Prins M, Buller HR. Randomized trial of the effect of the low molecular weight heparin nadroparin on survival in patients with cancer. J Clin Oncol. 2011 May 20;29(15):2071-6. doi: 10.1200/JCO.2010.31.9293. Epub 2011 Apr 18. PMID 21502549
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: FRX106365 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FRX106365 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FRX106365 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: FRX106365 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: FRX106365 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FRX106365 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FRX106365 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register